CLINICAL TRIAL: NCT04120779
Title: Study Protocol of the EMPOWER-SUSTAIN Project: A Pilot Randomised Controlled Trial of e-Health Intervention to Improve Patient Activation and Self-Management Behaviours Among Individuals With Metabolic Syndrome in Primary Care Setting
Brief Title: Study Protocol of the EMPOWER-SUSTAIN Project
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universiti Teknologi Mara (Other)
Collaborators: Ministry of Education, Malaysia (Other Government)
Responsible Party: Principal Investigator, Professor Dr. Anis Safura Ramli, Professor, Universiti Teknologi Mara
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: EMPOWER-SUSTAIN Project
Record Dates: First submitted 2019-10-04; First posted 2019-10-09 (Actual); Last update posted 2020-11-23 (Actual); Status verified 2020-11

CONDITIONS: Metabolic Syndrome
Keywords: e-health intervention; self-management; primary care; chronic care model
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Intervention Model Description: Pilot Randomised Controlled Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The EMPOWER-SUSTAIN e-Health Intervention (Experimental): The EMPOWER-SUSTAIN intervention is a multifaceted chronic disease management strategies based on the Chronic Care Model (CCM) and persuasive technology (PT) theory. It consists of training physicians and patients to use the EMPOWER-SUSTAIN web-based self-management intervention mobile apps, strengthening patient-physician relationship and reinforcing the use of relevant clinical practice guidelines for management and prescribing.
  Interventions: Device: The EMPOWER-SUSTAIN e-Health Self-Management Intervention
- Control (No Intervention): The control group will continue to receive usual care at the university primary care clinic. They will be given the EMPOWER-SUSTAIN Global CV Risks Self-Management Booklet©, as this is considered as usual care at the university primary care clinic. The EMPOWER-SUSTAIN web-based self-management tool will be made available to the control group at the end of the study. During the course of the study, there will be no limit to the number of clinic visits that a patient is allowed to make in either the intervention or control groups.

INTERVENTIONS:
Device: The EMPOWER-SUSTAIN e-Health Self-Management Intervention — Multifaceted chronic disease management strategies involving web-based self-management intervention mobile apps based on chronic care model and persuasive technology theory to improve patient activation and self-management behaviours among patients with metabolic syndrome.
  Arms: The EMPOWER-SUSTAIN e-Health Intervention

SUMMARY:
A pilot randomised controlled trial will be conducted in UiTM Primary Care Clinic, Selayang Campus, Selangor, Malaysia. A total of 232 patients with Metabolic Syndrome (MetS) will be recruited; 116 will be randomised to receive the EMPOWER-SUSTAIN intervention for 6 months and another 116 patients will continue with usual care. The EMPOWER-SUSTAIN intervention is a multifaceted chronic disease management strategies based on the Chronic Care Model (CCM) and persuasive technology theory. It consists of training physicians and patients to use the EMPOWER-SUSTAIN web-based self-management intervention mobile apps, strengthening patient-physician relationship and reinforcing the use of relevant clinical practice guidelines for management and prescribing. The primary outcome is the mean change in patient activation score using the Patient Activation Measure short form Malay version (PAM-13-M) questionnaire. The secondary outcomes include the change in patients' physical activity level, eating behavior, patients' perception on chronic illness care, satisfaction in physician-patient interaction and perceived absolute 10-year cardiovascular disease (CVD) risk.

DETAILED DESCRIPTION:
Study Design:

This is a pilot randomised controlled trial. The overall duration of the study is one year, and the duration of the intervention is 6 months. Blinding is not possible due to the nature and complexity of the intervention. The reporting of this paper is done in accordance with the SPIRIT 2013 guidance for protocols of clinical trials and the CONSORT checklist for pilot and feasibility trials. Figure 1 shows the EMPOWER-SUSTAIN CONSORT Flow Diagram.

Study Population:

The study population will comprise of individuals who are diagnosed with Metabolic Syndrome (MetS) according to the Joint Interim Statement (JIS) on MetS definition, 2009 by the International Diabetes Federation Task Force on Epidemiology and Prevention; National Heart, Lung, and Blood Institute; American Heart Association; World Heart Federation; International Atherosclerosis Society; and International Association for the Study of Obesity.

According to the JIS definition, MetS is defined by the presence of at least 3 out of 5 of the following risk factors:

I. Waist Circumference (WC): M ≥ 90 cm F ≥ 80 cm (South Asian cut-points) II. Blood Pressure (BP): Systolic BP ≥ 130 and/or diastolic BP ≥ 85 mmHg or on treatment for hypertension (HPT) III. Fasting Blood Glucose (FBG): ≥ 5.6 mmol/L or on treatment for elevated glucose IV. Triglycerides (TG): ≥ 1.7 mmol/L or on treatment for TG V. High density lipoprotein cholesterol (HDL-c): Male < 1.0 mmol/L, Female < 1.3 mmol/L; or on treatment for HDL-c

Patient Recruitment:

Consecutive patients who attend the UiTM Primary Care Clinic during the recruitment period will be approached, given the patient information sheet about the study and invited to participate. Those who are willing to participate will be interviewed and screened by the investigators to identify eligibility based on the inclusion and exclusion criteria. Written informed consent will be obtained from those who are eligible and they will be recruited into the study.

Physician Recruitment:

All primary care physician (PCP) who are practicing at the university primary care clinic will be invited to participate in the study. To be eligible, the following criteria must be met:

1. have one or more years of working experience in a primary care setting
2. must be keen to participate in the study
3. willing to deliver the EMPOWER-SUSTAIN e-Health Intervention to patients with MetS

The Intervention:

The EMPOWER-SUSTAIN Self-Management e-Health Intervention is a complex intervention involving multifaceted components based on the CCM and persuasive technology approach. A comprehensive review of the literature was conducted to identify the crucial components of e-health intervention that could improve patient activation and self-management behaviours. The EMPOWER-SUSTAIN intervention is a multifaceted chronic disease management strategies based on the CCM and persuasive technology theory. It consists of training physicians and patients to use the EMPOWER-SUSTAIN web-based self-management intervention mobile apps, strengthening patient-physician relationship and reinforcing the use of relevant clinical practice guidelines for management and prescribing.

Conduct of the EMPOWER-SUSTAIN Workshop:

Prior to the intervention, PCP and patient with MetS in the intervention arm will be trained on the EMPOWER-SUSTAIN web-based desktop and mobile applications utilisation in the EMPOWER-SUSTAIN Workshop.

Delivery of the Intervention:

The EMPOWER-SUSTAIN Self-Management e-Health Intervention will be professionally delivered to the individual patient by the PCP. Patients will also be given the EMPOWER-SUSTAIN Global CV Risks Self-Management Booklet©. Follow-up care by the PCP will be arranged at baseline, 3-month and 6-month. At baseline, PCP assisted by a nurse, will go through each section with the patient and will ensure that information recorded in all sections is complete. PCP will discuss self-management progress and goals using this tool with the patient at each follow-up visit. Patients will be able to review their progress at home and use the tool to aid self-management of their MetS e.g. self-monitoring of their weight, BP and blood glucose, recording of their physical activity and diet.

Monitoring the Intervention:

During the 6-month intervention period, patients are required to utilize the EMPOWER-SUSTAIN web-based self-management tool for a cumulative period of two hours duration, and be seen at least once by the PCP for follow-up care. A separate web interface will be created for PCP to monitor patient's log-in frequency and duration of utilisation of the tool. Patients who do not comply with the utilization and follow-up requirements will be considered as lost to follow-up. Patients who are lost to follow-up or who withdraw from the trial will not be replaced. Analysis will be by intention to treat. There is no limit to the number of clinic visit a patient is allowed to make in either arm during the course of the study.

Study Tools:

1. Patient Activation Measure short form - Malay version (PAM-13-M) questionnaire
2. International Physical Activity Questionnaire - Malay version (IPAQ-M)
3. Dutch Eating Behaviour Questionnaire - Malay version (DEBQ-M)
4. Patients Assessment of Chronic Illness Care - Malay version (PACIC-M) questionnaire
5. Skala Kepuasan Interaksi Perubatan (SKIP-11) questionnaire
6. Perceived absolute 10-year CVD risk and the actual calculated risk by Framingham Risk Score (FRS) General CVD risk prediction chart.

Sample Size Determination:

Sample size is calculated using Power and Sample Size Calculation software version 3.1.2, 2014 based on the findings of a randomised controlled trial evaluating the effects of a web-based self-management intervention for adults with chronic conditions on patient activation scores, measured by the PAM-13 questionnaire. In the intervention group, the mean patient activation score at baseline was 65.33 and the mean score after the intervention was 71.30 (mean difference of 5.97 ± 9.70, t57 = 4.683, P < 0.001). Whereas, in the control group, the mean patient activation score at baseline was 66.89 and the mean score at the end of the study period was 68.93 (mean difference of 2.04 ± 10.01, t67 = 1.677, P= 0.10). Therefore, the mean difference between the two groups was 3.93.

Based on this assumption, a sample size of 97 participants per group is sufficient to detect mean difference of δ = 3.93 in the patient activation score between the two groups, with a standard deviation of σ = 9.70 using two-tailed t-test of difference between means with 80% power (power = 0.8), 5% level of significance (α = 0.05) and sample size ratio of 1:1 between the two groups (m =1). After considering a drop-out rate of 20%, the sample size required is 116 participants per group, giving a total of 232 patients to be recruited for this study.

Randomisation:

Randomisation of patients to either the EMPOWER-SUSTAIN Self-Management e-Health Intervention (I) or usual care (C) will be done using Randomised Block Design. Random allocation will be made in order to keep the sizes of the group similar. In this study, the block randomisation size will be 4 times the number of treatment arms i.e. block size of 2 by 2. With two treatment arms of the EMPOWER-SUSTAIN Self-Management e-Health Intervention (I) or usual care (C), the possible treatment allocations within each block will be as follows: IICC, ICIC, ICCI, CCII, CICI, CIIC.

Data Management:

Data will be checked before the end of each consultation to ensure the completeness of the questionnaire. If any missing data is found, the patients will be contacted again through the telephone. Raw data obtained will be entered in Excel and SPSS version 24.

Feasibility Outcomes:

Process evaluation to assess the integrity of the trial protocol will be conducted. Data to assess the integrity of the randomised controlled trial protocol will be collected. This include recruitment rate, methods of randomisation, retention rate, selection of primary/secondary outcome measures, sample size calculation, whether the intervention is delivered as intended and methods of statistical analysis to evaluate the potential effectiveness.

Statistical Analysis Plan:

The analysis will be conducted using SPSS version 24

Descriptive Analysis:

The frequency distribution, a measure of central tendency and dispersion will be produced. For the continuous data, it will be presented by mean and standard deviation or median based on the normality of the data. For the categorical data, it will be presented by absolute number and their corresponding percentages.

Effectiveness Analysis:

Intention to Treat (ITT) analysis will be applied to measure the potential effectiveness of the EMPOWER-SUSTAIN Self-Management e-Health Intervention on the primary and secondary outcome measures based on the initial treatment assignment. The mixed model repeated measure analysis of variance (ANOVA) will be carried out to evaluate the potential effectiveness i.e. to compare the mean changes in patient activation, physical activity, diet, patients' chronic illness care and physician-patient interaction satisfaction scores, perceived absolute 10-year CVD risk within and between the intervention and control groups at baseline and 6-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with MetS according to the JIS definition
* have received follow-up care for MetS at the university primary care clinic at least twice in the last one year
* have regular access to the internet
* perceive that they have basic skills to use the web and smart mobile phone
* are able to read and understand written English or Malay

Exclusion Criteria:

* type 1 diabetes mellitus
* receiving renal dialysis
* resented with severe hypertension (Systolic BP > 180 mmHg and/or Diastolic BP > 110 mmHg) at recruitment
* diagnosed with conditions resulting in secondary hypertension
* diagnosed with circulatory disorders requiring referral to secondary care over the last one year and during the course of the study
* receiving shared care at primary and secondary care centres for cardiovascular diseases
* receiving chemotherapy/ radiotherapy or palliative care
* diagnosed with a psychiatric illness such as schizophrenia, bipolar disorder, major depression
* diagnosed with cognitive impairment such as dementia
* pregnant
* enrolled in another intervention study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 232 (Estimated)
Dates: Start 2021-03-01 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
The mean change in patient activation score using the Patient Activation Measure short form Malay version (PAM 13-M) questionnaire. | 6 months
  The PAM-13 consists of 13 items measuring patients' self-reported knowledge, skills and confidence for self-management. Each item is scored on a Likert scale of 1-5. The instrument reflects the 4 stages of activation in a progressing difficulty of the items: level 1 (patients believe that their role is important), level 2 (patients have confidence and knowledge to take action), level 3 (taking action) and level 4 (staying on course under stress). According to the scoring guidelines, the raw scores are transformed through natural logarithm to achieve a better expression of the relative distance between the scores. Then, items are transformed to a standardized metric ranging from 0 to 100 (0 = lower activation; 100 = highest activation). The score is calculated by summing up the raw scores and mapping up the sum onto a scale of 0-100. A higher score of PAM-13 indicates a high level of patients activation.

SECONDARY OUTCOMES:
Change in physical activity level using the International Physical Activity Questionnaire short form Malay version (IPAQ-M) | 6 months
  The IPAQ-M short version comprises of 12 items, covering vigorous, moderate, walking, sitting and sleeping activities. Patients are required to report the activities performed during the last seven days and to include only activities that lasted 10 minutes or more per session. IPAQ will be scored according to its scoring protocol. Continuous score will be expressed as Metabolic Equivalent Task (MET)-minutes per week: MET level x minutes of activity/day x days per week. The scores will then be categorised into 'Low', 'Moderate' and 'Vigorous' physical activity level, in accordance to the Malaysian Clinical Practice Guideline on Primary and Secondary Prevention of Cardiovascular Disease 2017.
Change in eating behaviour will be measured by the Dutch Eating Behaviour Questionnaire - Malay version (DEBQ-M) | 6 months
  The DEBQ-M contains 33 items to measure emotional, external, and restrained eating behaviours. Emotional eating is assessed by 13 items, whereas external and restrained eating behaviours are assessed by 10 items each. The questions that assess the three different behaviours appear in random order in the questionnaire and are answered according to the Likert scale with a scoring system identified as follows: 1 = never, 2 = rarely, 3 = sometimes, 4 = often, and 5 = very often. There are three sub-scales in the instrument. For each subscale, the score is added and divided by the number of items in the sub-scale to obtain the average score for emotional, external and restrained eating for a person.
Change in patients' perceptions and experiences of receiving care for chronic conditions will be measured by the Patients Assessment of Chronic Illness Care Malay version (PACIC-M) questionnaire | 6 months
  The PACIC-M questionnaire consists of 20-item patient self-reported instrument to assess the extent to which patients with chronic disease receive care that aligns with the Chronic Care Model. It measures care that is patient-centred, proactive and planned, which includes collaborative goal setting, problem-solving and follow-up support. Each item is scored on a 5-point Likert scale with 1 being 'no' or 'never' and 5 being 'yes' or 'always'. The higher the score, the more aligned is the perceived care to CCM.
Change in patient-physician satisfaction will be measured by the the Skala Kepuasan Interaksi Perubatan (SKIP 11) questionnaire | 6 months
  SKIP-11 is the translated and validated Malay version of the Medical Interview Satisfaction Scale (MISS-21). It consists of 11 questions representing 3 subdomains of physician-patients interaction satisfaction: 'Distress relief', 'Rapport' and 'Interaction Outcome'. All 11 items are scored using a 5-point Likert scale. Each response will be added together to give a total score within the range of 11 (minimum) and 55 (maximum). Total score for each subdomain is also calculated and analysed where the minimum and maximum score is determined by the number of items present in each subdomain. The levels of satisfaction will be determined by the proximity of the score to either the minimum or maximum score for each subdomain. The closer proximity of the score to the maximum score will reflect good satisfaction level and vice versa.
Change in the accuracy of the Perceived Absolute 10-year CVD Risk | 6 months
  The accuracy of the CVD risk perception will be measured by the absolute difference between the perceived absolute10-year CV risk and the actual calculated risk by FRS General CVD risk prediction chart. The absolute difference will be inversely related i.e. the lower is the absolute difference, the more accurate is the patients' CVD risk perception.

CONTACTS AND LOCATIONS:
Overall Officials: Anis S Ramli, Prof. Dr., Principal Investigator — Institute of Pathology, Laboratory and Forensic Medicine (I-PPerForM)

IPD SHARING:
Plan to Share IPD: No
Data will be kept at the Institute of Pathology, Laboratory and Forensic Medicine (I-PPerForM), Universiti Teknologi MARA (UiTM), Sungai Buloh Campus, Jalan Hospital, 47000 Sungai Buloh, Selangor, Malaysia. Data can be shared upon request and is subjected to the data protection regulations.

REFERENCES:
- [Background] Chan AW, Tetzlaff JM, Gotzsche PC, Altman DG, Mann H, Berlin JA, Dickersin K, Hrobjartsson A, Schulz KF, Parulekar WR, Krleza-Jeric K, Laupacis A, Moher D. SPIRIT 2013 explanation and elaboration: guidance for protocols of clinical trials. BMJ. 2013 Jan 8;346:e7586. doi: 10.1136/bmj.e7586. PMID 23303884
- [Background] Eldridge SM, Chan CL, Campbell MJ, Bond CM, Hopewell S, Thabane L, Lancaster GA; PAFS consensus group. CONSORT 2010 statement: extension to randomised pilot and feasibility trials. BMJ. 2016 Oct 24;355:i5239. doi: 10.1136/bmj.i5239. PMID 27777223
- [Background] Alberti KG, Eckel RH, Grundy SM, Zimmet PZ, Cleeman JI, Donato KA, Fruchart JC, James WP, Loria CM, Smith SC Jr; International Diabetes Federation Task Force on Epidemiology and Prevention; Hational Heart, Lung, and Blood Institute; American Heart Association; World Heart Federation; International Atherosclerosis Society; International Association for the Study of Obesity. Harmonizing the metabolic syndrome: a joint interim statement of the International Diabetes Federation Task Force on Epidemiology and Prevention; National Heart, Lung, and Blood Institute; American Heart Association; World Heart Federation; International Atherosclerosis Society; and International Association for the Study of Obesity. Circulation. 2009 Oct 20;120(16):1640-5. doi: 10.1161/CIRCULATIONAHA.109.192644. Epub 2009 Oct 5. PMID 19805654
- [Background] Hibbard JH, Mahoney ER, Stockard J, Tusler M. Development and testing of a short form of the patient activation measure. Health Serv Res. 2005 Dec;40(6 Pt 1):1918-30. doi: 10.1111/j.1475-6773.2005.00438.x. PMID 16336556
- [Background] Chu AH, Moy FM. Reliability and validity of the Malay International Physical Activity Questionnaire (IPAQ-M) among a Malay population in Malaysia. Asia Pac J Public Health. 2015 Mar;27(2):NP2381-9. doi: 10.1177/1010539512444120. Epub 2012 May 16. PMID 22593217
- [Background] Subramaniam K, Low WY, Chinna K, Chin KF, Krishnaswamy S. Psychometric Properties of the Malay Version of the Dutch Eating Behaviour Questionnaire (DEBQ) in a Sample of Malaysian Adults Attending a Health Care Facility. Malays J Med Sci. 2017 Aug;24(4):64-73. doi: 10.21315/mjms2017.24.4.8. Epub 2017 Aug 18. PMID 28951691
- [Background] Abdul-Razak S, Ramli AS, Badlishah-Sham SF, Haniff J; EMPOWER-PAR Investigators. Validity and reliability of the patient assessment on chronic illness care (PACIC) questionnaire: the Malay version. BMC Fam Pract. 2018 Jul 19;19(1):119. doi: 10.1186/s12875-018-0807-5. PMID 30025525
- [Background] Abd Aziz A, Izyan Farhana Nordin N, Mohd Noor N, Bachok N, Nor Ismalina Isa S. Psychometric properties of the 'Skala Kepuasan Interaksi Perubatan-11' to measure patient satisfaction with physician-patient interaction in Malaysia. Fam Pract. 2014 Apr;31(2):236-44. doi: 10.1093/fampra/cmt062. Epub 2013 Dec 6. PMID 24317538
- [Background] Frijling BD, Lobo CM, Keus IM, Jenks KM, Akkermans RP, Hulscher ME, Prins A, van der Wouden JC, Grol RP. Perceptions of cardiovascular risk among patients with hypertension or diabetes. Patient Educ Couns. 2004 Jan;52(1):47-53. doi: 10.1016/s0738-3991(02)00248-3. PMID 14729290
- [Background] Solomon M, Wagner SL, Goes J. Effects of a Web-based intervention for adults with chronic conditions on patient activation: online randomized controlled trial. J Med Internet Res. 2012 Feb 21;14(1):e32. doi: 10.2196/jmir.1924. PMID 22353433
- [Derived] Palmer MJ, Machiyama K, Woodd S, Gubijev A, Barnard S, Russell S, Perel P, Free C. Mobile phone-based interventions for improving adherence to medication prescribed for the primary prevention of cardiovascular disease in adults. Cochrane Database Syst Rev. 2021 Mar 26;3(3):CD012675. doi: 10.1002/14651858.CD012675.pub3. PMID 33769555
- [Derived] Daud MH, Ramli AS, Abdul-Razak S, Isa MR, Yusoff FH, Baharudin N, Mohamed-Yassin MS, Badlishah-Sham SF, Nikmat AW, Jamil N, Mohd-Nawawi H. The EMPOWER-SUSTAIN e-Health Intervention to improve patient activation and self-management behaviours among individuals with Metabolic Syndrome in primary care: study protocol for a pilot randomised controlled trial. Trials. 2020 Apr 5;21(1):311. doi: 10.1186/s13063-020-04237-x. PMID 32248825